CLINICAL TRIAL: NCT06803511
Title: Investigating the Relationship Between Dietary Acid Load and Oral Health-Related Quality of Life in Adolescents
Brief Title: Dietary Acid Load and Oral Health Quality in Adolescents
Status: Completed | Type: Observational
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Principal Investigator, Emine Elibol, Assist. Prof., Ankara Yildirim Beyazıt University
Other Study IDs: AYBUELİBOL007
Record Dates: First submitted 2025-01-27; First posted 2025-01-31 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2024-12

CONDITIONS: Adolescent
Keywords: Dietary acid load; oral health; quality of life; adolescents

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Adolescents: This study investigates the link between dietary acid load and oral health-related quality of life in 374 high school students (226 females, 148 males). Participants completed a demographic questionnaire, the OHIP-14 scale, and provided 24-hour dietary recalls. Dietary acid load was assessed using PRAL and NEAP calculations. Data analysis was performed with SPSS 24 to explore the impact of diet composition on adolescents' oral health.

SUMMARY:
This study investigates the link between dietary acid load and oral health-related quality of life in 374 high school students (226 females, 148 males). Participants completed a demographic questionnaire, the OHIP-14 scale, and provided 24-hour dietary recalls. Dietary acid load was assessed using PRAL and NEAP calculations. Data analysis was performed with SPSS 24 to explore the impact of diet composition on adolescents' oral health.

DETAILED DESCRIPTION:
Introduction: Oral health plays a crucial role in the psychological and physical development of children and adolescents. The composition of the diet consumed significantly affects oral health.

Objective: This study aimed to examine the relationship between dietary acid load and oral health-related quality of life in adolescents.

Method: A total of 374 high school students (226 females, 148 males) participated in the study. Adolescents completed a demographic questionnaire and the Oral Health Impact Profile-14 (OHIP-14) scale, and 24-hour retrospective food consumption records were collected. Dietary acid load was assessed by calculating potential renal acid load (PRAL) and net endogenous acid production (NEAP) based on macronutrient and micronutrient intake from food records. Data analysis was conducted using the SPSS 24 software package.

ELIGIBILITY:
Inclusion Criteria:

* 14-18 ages

Exclusion Criteria:

* those with diagnosed eating disorders
* those with diagnosed psychiatric
* those with diagnosed cancer

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Community sample in Türkiye
Sampling Method: Non-Probability Sample
Enrollment: 374 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-05-15 (Actual); Study Completion 2024-06-15 (Actual)

PRIMARY OUTCOMES:
Oral Health Impact Profile-14 Score | Baseline
  This scale was used to assess the quality of life related to oral health and how oral health affects overall quality of life and general health.
  The scale consists of 14 items with 5-point Likert-type questions (each option ranging from 0 to 4 points) and was designed using a five-choice scaling method. It was concluded that as the total score increased, the severity of the problem also increased, leading to a decrease in quality of life.
Calculation of Dietary Acid Load | Baseline
  Dietary acid load (DAL), potential renal acid load (PRAL), and net endogenous acid production (NEAP) were calculated based on the 24 hours food consumption record The formula for PRAL is as follows:
  PRAL (mEq/day) = 0.4888 x protein (g/day) +0.0366 x phosphorus (mg/day)-0.0205 x potassium (mg/day) - 0.0125 x calcium (mg/day) - 0.0263 x magnesium (mg/day) NEAP (mEq/day) = [54.5 x protein (g/day) / potassium (mEq/day)] - 10.2 High and positive PRAL and NEAP values indicate a high dietary acid load.

SECONDARY OUTCOMES:
Sociodemographic characteristics | Baseline
  Sociodemographic characteristics will be assessed using a structured questionnaire developed by the researchers. The questionnaire will include items measuring age, gender, education level, and income status. The results will be presented as numbers and percentages for each characteristic.
Body Mass Index (BMI) | Baseline
  Kilograms per square meter (kg/m2)
Height | Baseline
  Height in cm
Body weight | Baseline
  Body weight in kg

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Yıldırım Beyazıt University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No